CLINICAL TRIAL: NCT00622271
Title: Adjustment and Self-Management Intervention Groups for Adolescents With Type 1 Diabetes Mellitus and Their Parents.
Brief Title: Intervention Groups for Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Jessica C. Kichler, Psychologist, Children's Hospital and Health System Foundation, Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTP1
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Adolescents and Families; Group Therapy Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wait List Control (Other): Patients and their families will be enrolled into either a treatment group or a wait list control (WLC) group to receive the group therapy intervention.
  Interventions: Behavioral: Group Therapy

INTERVENTIONS:
Behavioral: Group Therapy — Self-management Group Protocol: The parent sessions will be structured by general topic area, but teaching of clinical and behavioral information will be derived from questions and problems posed by the group in order to actively meet the needs and concerns of participants. The parent sessions will be an interactive process of eliciting concerns and questions, presenting information to address those questions, and following up with a discussion to review concerns and strategies to address the behavioral aspects of the issues. The child sessions will be activity focused, with hands-on opportunities to practice the skills being taught.

SUMMARY:
The purpose of this study is to utilize a group therapy adjustment and coping program at the Children's Hospital of Wisconsin with patients who have Type 1 Diabetes Mellitus (T1DM) and their parents within a "typical" clinical condition of patients who have been referred for outpatient therapy services. To extend the previous literature on these types of peer and family-based groups to include survey data as well as provider ratings, medical data, and add retrospective and prospective data from baseline enrollment. To aid in establishing this group therapy methodology as a "promising" evidence-based intervention within a population of youths with T1DM and their families. The specific aim of this project is to enroll patients and their families into either a treatment group or a wait list control group to receive the group intervention to determine the impact of this peer and family-based group on improving adjustment, coping, and functioning within diabetes.

DETAILED DESCRIPTION:
A total sample size of approximately 40 youth participants and their parents (4 x 6-10) in two waves will be recruited. More specifically, there will be a treatment group (n = 6-10) and a wait list control group (n = 6-10) who participate in the first wave and another treatment group (n = 6-10) and wait list control group (n = 6-10) in the second wave. This number was chosen on the basis of including an adequate number of participants to appropriately demonstrate the effectiveness of the protocol within a clinical setting, the recommendations to conduct group therapy in cohorts of 6-10 to be the most effective clinically, and the pragmatics of participant availability based on the referral rates from the Diabetes Clinic in the past for mental health treatment. In addition, having 6-10 participants will allow for some participant attrition without impacting the effectiveness of the group therapy.

All families with an eligible participant, an adolescent between the ages of 13-17 years old with T1DM who is seen at the Children's Hospital of Wisconsin Diabetes clinic, will be recruited by diabetes providers and study researchers in the Diabetes Clinics and education classes, and from referrals to the Child and Adolescent Psychiatry and Behavioral Medicine Center Clinic. They will be given a flyer describing the study. Families will contact the intake coordinators at the Child and Adolescent Psychiatry and Behavioral Medicine Center to receive a phone intake and be screened for appropriateness of their participation in the group therapy. An insurance verification will also be completed to determine insurance coverage for participating in the group. If a family is not eligible or declines to participate in the group therapy research, they will be referred for individual therapy. For those participants who do qualify and agree verbally to participate, plans will be made for the family to participate in an intake session. At that initial intake visit, if they remain interested in participating in this study, they will be randomly assigned to the treatment group or the WLC group per the CONSORT Guidelines (Moher et al., 2001). Once they have arrived for their intake appointment in the Child and Adolescent Psychiatry and Behavioral Medicine Center, the parents and adolescents will be asked to give informed consent/assent for both the clinical and research aspects of the group therapy. They will then complete the questionnaires before their intake session. In addition, participants will be recruited through an advertisement in the Children's Hospital of Wisconsin diabetes newsletters/mailings as well as postings of the advertisement flyer and recruitment in the Diabetes Clinic.

Following parental consent and adolescent assent, the parents will complete standardized measures of general demographic information, general psychosocial functioning (e.g., quality of life, emotional and behavioral functioning of their child, parent stress, health-related family impact), and diabetes-related functioning (e.g., adherence, readiness to change behaviors, responsibility, health-related quality of life, health satisfaction). The adolescents will be asked to complete measures of general demographic information, general psychosocial functioning (e.g., quality of life, and emotional and behavioral functioning), and diabetes-related functioning (e.g., adherence, readiness to change behaviors, responsibility, health-related quality of life). For the treatment group, these measures will be given again at post-treatment and then at 4 months after baseline. For the WLC group, these measures will be given again at the initiation of group therapy, post-treatment, and 4 months after starting group treatment. (Please see attached schedule of assessments for reference). The length of time to complete these questionnaires is estimated to be around 45 minutes.

In addition to the self-report measures, each participant's medical record will be reviewed for information for the 6 months prior to baseline and the 6 months after the start of group therapy to obtain height, weight Tanner scores, hospital admissions related to diabetes, ER visits related to T1DM, outpatient diabetes clinic visits, severity of diabetes ketoacidosis (DKA) admissions through pH and HCO3 mEq/L lab work, Hemoglobin A1c levels, categorical ratings of diabetes status, and absentee rates at school from the outpatient clinic notes during the participation time period. The duration and type of diabetes reported by parents will be verified during the medical record review. We will track inpatient and outpatient hospital charges for diabetes that occur in the CHW system during the participation time frame.

Participants will be treated as outpatient clinic patients and will be responsible for all costs associated with care, including group therapy charges. Funds are not available for payment of diabetes self-management education (DSME) fees, clinic fees, lab fees, hospitalization or reimbursement of participants. Any medical or mental health costs outside of the clinical and research materials (e.g., surveys, copies, and supplies for group therapy) during the intervention will be the responsibility of the participant's family or third party insurer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been referred for outpatient therapy services will be included if they have Type 1 Diabetes and are 13-17 years of age.

Exclusion Criteria:

* Potential participants will be excluded if they have the following co-existing diagnoses: mental retardation, pervasive developmental disorders, substance abuse, eating disorders, psychosis, other acute psychiatric or medical needs, such as suicidality.
* Potential participants will be excluded if they are not fluent in the English language.
* If a family is not eligible or declines to participate in the group therapy research, they will be referred for individual therapy.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Enroll patients and their families into either a treatment group or a wait list control (WLC) group to determine the impact of a peer and family-based group intervention on improving adjustment, coping, and functioning among adolescents with diabetes. | Baseline, end of treatment, 4 months post-treatment, and 6 months post treatment

SECONDARY OUTCOMES:
Cost-effectiveness will be demonstrated through decreased health care utilization (e.g., emergency room visits, extra outpatient visits, and inpatient hospitalizations). | 6 months prior to initiating treatment and 6 months after initiating treatment
Diabetes-related medical improvements from baseline to post-treatment and maintained at 4 months and 6 months post-treatment. | baseline, post-treatment, 4 months and 6 months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica C Kichler, Ph.D., Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin Child and Adolescent Psychiatry and Behavioral Medicine Center and the Diabetes Clinic, Milwaukee, Wisconsin, United States